CLINICAL TRIAL: NCT05146973
Title: A Single Arm, Phase 2 Trial of External Beam Radiation Therapy (EBRT) in Combination With 177Lu-DOTA-TLX591-CHO in Patients With Biochemically Recurrent Oligometastatic, Prostate Specific Membrane Antigen-Expressing Prostate Cancer
Brief Title: External Beam Therapy With Theranostic Radioligand Therapy for Oligometastatic Prostate Cancer (ProstACT TARGET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProstACT TARGET
Record Dates: First submitted 2021-11-25; First posted 2021-12-07 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single administration of 177Lu-DOTA-TLX591 (Experimental): Two single IV infusions of 76 mCi (2.8 GBq) each (equivalent to a 45 mCi/m2 administered activity in a standard 1.7m2 individual) of 177Lu-DOTA-TLX591, given 14 days apart.
  Interventions: Biological: 177Lu-DOTA-TLX591

INTERVENTIONS:
Biological: 177Lu-DOTA-TLX591 — TLX591, a monoclonal antibody conjugated with a DOTA chelator and radiolabelled with 177Lu (177Lu-DOTA-TLX591)

SUMMARY:
This is a phase II trial to evaluate the therapeutic efficacy of a radiolabelled PSMA-targeting antibody, 177Lu-TLX591, given in combination with external beam radiation therapy (EBRT) in patients with biochemically recurrent, oligometastatic, PSMA-expressing prostate cancer. TLX591 is being developed as a PSMA-targeting antibody to be radiolabelled with a therapeutic radioisotope for the treatment of PSMA-expressing tumours.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male, aged ≥ 18 years
* Estimated life expectancy of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) score 0 - 2
* Biopsy proven prostate adenocarcinoma with Gleason Score 7 or more at primary presentation
* Previous Radical Prostatectomy (RP) with curative intent (+/- post-operative radiotherapy to prostate bed)
* Biochemical relapse, as defined by EAU-ESTRO-SIOG Guidelines (serum PSA > 0.2 ng/mL, confirmed by repeat measurements)
* PSMA-ligand avid pelvic nodal disease on PSMA-ligand PET/CT, with visualised disease confined to the pelvis with or without evidence of PSMA-avid disease in the prostate bed
* At least one pelvic nodal lesion ≥ 5 mm in the greatest dimension. SUVmax > 9 in enlarged nodes; SUVmax > 3 in nodes 5 mm or less
* Oligometastatic disease as defined by ≤ 5 metastatic lymph nodes
* Metastatic lymph nodes not beyond the aortic bifurcation
* Non-castrate levels of testosterone (> 20 ng/dL)
* Chemotherapy naïve
* Adequate renal function: Cr Cl ≥ 40 mL/min (determined by Cockcroft-Gault formula)
* Adequate bone marrow function: Hb > 90 g/L; platelets > 100 x 109/L; neutrophils > 1.5 x 109/L
* Adequate liver function: bilirubin < 1.5 x upper limit of normal (ULN); AST, ALT, ALP < 2 x ULN; albumin > 30 g/L
* Willing and able to comply with all trial requirements, including all treatments and pre- and post-treatment assessments
* Able to commence treatment within 28 days of enrolment

Exclusion Criteria:

* Previous external beam radiotherapy to pelvis for other malignancies or medical conditions (except for post-operative prostate bed radiotherapy for prostate cancer)
* Androgen deprivation therapy within 12 months of trial screening
* Known androgen deficiency
* Bone or visceral metastases
* Lymph node metastases above the aortic bifurcation
* Contraindications to pelvic irradiation as determined by Investigator (e.g., chronic inflammatory bowel disease)
* At increased risk of haemorrhage, or recent history of a thrombotic event (e.g., Deep Vein Thrombosis [DVT]/Pulmonary Embolism [PE]) and/or are using long-term anti-coagulant or anti-platelet agents)
* Known hypersensitivity to any isotope of lutetium (Lu) in any chemical form, or any isotope used in PSMA imaging
* Contraindication to intravenous contrast
* Evidence of urinary tract stricture, or significant urinary/faecal incontinence Presence of active infection at time of screening, or history of serious infection within the previous 4 weeks
* History of any malignancy other than prostate cancer within 5 years of enrolment (excluding localised non-melanoma skin cancers)
* Any uncontrolled significant medical, psychiatric, or surgical condition (e.g., active infection, unstable angina pectoris, cardiac arrhythmia, poorly controlled type 2 diabetes, uncontrolled congestive heart failure, pulmonary disease), or laboratory findings that, in the opinion of the Investigator, may jeopardise the participant's safety or that would limit compliance with the treatment and assessment requirements of the trial
* Any cognitive impairment or other condition that may render the participant unable to adequately understand the requirements, nature, and possible consequences of the trial.
* Intention to father children within a timeframe corresponding with the duration of the allocated treatment regime plus 12 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
To determine Prostate Specific Antigen Progression Free Survival (PSA PFS) | Through study completion, up to 2 years
  The time from enrolment to time of PSA increase greater than 25%

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - GenesisCare North Shore, St Leonards, New South Wales
  - GenesisCare Murdoch, Perth, Western Australia
  - GenesisCare St Andrews, Adelaide
  - GenesisCare Tugun, Tugun

IPD SHARING:
Plan to Share IPD: No